CLINICAL TRIAL: NCT02118064
Title: A Multinational, Multicenter, Open-label, Single-arm, Phase II Study of G17DT Immunogen in Combination With Irinotecan in Metastatic Colorectal Carcinoma Refractory to Previous Irinotecan-based Chemotherapy.
Brief Title: Phase II Study to Evaluate G17DT in Combination With Irinotecan in Patients With Colorectal Carcinoma
Acronym: CC6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC6
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer
Keywords: G17DT; irinotecan; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

ARMS (1):
- G17DT-Irinotecan (Experimental): 500µg dose of G17DT intramuscular injection in combination with 125 mg/m^2 intravenous infusion of Irinotecan over 90 minutes.
  Interventions: Biological: G17DT-Irinotecan

INTERVENTIONS:
Biological: G17DT-Irinotecan — 500µg dose of G17DT intramuscular injection in combination with 125 mg/m^2 intravenous infusion of Irinotecan over 90 minutes.

SUMMARY:
This study was designed to evaluate the ability for G17DT to slow or arrest tumor growth in patients with refractory colon cancer who had been previously treated with an Irinotecan-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed cancer of the colon or rectum or both and objective evidence of distant metastases
* Have measurable disease
* Have previously been treated with an irinotecan based chemotherapy
* Have progressive metastatic disease after an irinotecan containing chemotherapy regimen (alone or in combination) for metastatic colorectal cancer
* Be at least 18 years of age
* Have laboratory data as specified below:

  * Aspartate aminotransferase (AST) and ALT less than 2.5 times upper limit of normal
  * Bilirubin less than 1.5 mg/dL (SI units, 25.65 mol/L)
  * Creatinine less than 1.5 mg/dL (SI units, 132 mol/L)
  * White blood cell (WBC) count greater than 3,000/mm3
  * Platelets greater than 100,000/mm3
  * Hemoglobin more than 9.5 g/dL (SI units, 5.9 mol/L)
  * International normalized ratio of prothrombin time less than 1.2, and activated partial thromboplastin time no more than 5 seconds above normal limits
* Have a life expectancy of at least 3 months
* Have a KPS score of 70 or greater
* Use contraceptive methods, if sexually active
* Have the ability to understand the requirements of the study, to provide written informed consent, agree to abide by the study restrictions, and agree to return for the required assessments

Exclusion Criteria:

* Be pregnant or nursing
* Have only symptomatic locally recurrent colorectal cancer
* Have had any active cancer in addition to metastatic colorectal cancer within the last 5 years except curatively treated nonmelanomatous skin cancer
* Have received any prior anticancer immunotherapy
* Have central nervous system metastasis, whether treated or not
* Have bone metastases as sole manifestation of metastatic colorectal cancer
* Have received chemotherapy within the previous 21 days
* Have had major surgery within 21 days
* Have immunodeficiency (primary or acquired)
* Have undergone bone marrow transplantation within the last year
* Require chronic administration of corticosteroids; inhaled corticosteroids for asthma and chronic obstructive pulmonary disease are allowed
* Use in the past 30 days or concomitant use of immunosuppressants, including systemic (i.e., oral or injected) corticosteroids
* Have participated in any clinical trial involving conventional or investigational drugs or devices within 21 days before G17DT irinotecan administration
* Have contraindication to irinotecan based therapy
* Have hypersensitivity to diphtheria toxoid
* Use in the past 14 days or chronic concomitant use of proton pump inhibitors
* Have uncontrolled serious cardiovascular or metabolic disease or any other uncontrolled serious medical or psychiatric illness
* Have any condition that is likely to detrimentally affect regular follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2001-03; Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Tumor response | up to 12 months
  Evaluate the effect of G17DT-Irinotecan combination therapy on tumor response assessed by magnetic resonance imaging or computed tomography.
Survival time | up to 12 months
  The vital status of patients was monitored until death or end of the study.
Number of Patients with Serious and Non-Serious Adverse Events | Up to 12 months
  Adverse events, defined as any event involving adverse reactions, illnesses with onset during the study, or exacerbations of pre-existing illnesses, were assessed at each visit.